CLINICAL TRIAL: NCT05268120
Title: MRSA Decolonization in Complicated Carriage - Cluster Randomized Trial
Brief Title: MRSA Decolonization in Complicated Carriage
Acronym: CLEANEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, acwestgeest, Principal investigator, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL79720.058.21
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-10

CONDITIONS: MRSA
MeSH Terms: interventions — Doxycycline; Trimethoprim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): doxycycline 200 mg q.d. - rifampicin 600mg b.i.d.
  Interventions: Drug: doxycycline 200 mg q.d. - rifampicin 600mg b.i.d.
- B (Active Comparator): trimethoprim 200mg b.i.d. - rifampicin 600mg b.i.d.
  Interventions: Drug: trimethoprim 200mg b.i.d. - rifampicin 600mg b.i.d.

INTERVENTIONS:
Drug: doxycycline 200 mg q.d. - rifampicin 600mg b.i.d. — Both first choice treatments in Dutch guideline for MRSA decolonization
  Arms: A
Drug: trimethoprim 200mg b.i.d. - rifampicin 600mg b.i.d. — Both first choice treatments in Dutch guideline for MRSA decolonization
  Arms: B

SUMMARY:
Multicenter open-label cluster randomized controlled trial determining the superiority of doxycycline-rifampicin compared to trimethoprim-rifampicin for the decolonization treatment of complicated MRSA carriership.

DETAILED DESCRIPTION:
Rationale: MRSA decolonization has proven to prevent infection and reduce transmission. It has yet remained undecided which combination of anti-staphylococcal agents is most effective in the treatment of complicated MRSA carriage. A recent cohort study showed the highest success rate of decolonization in patients treated with doxycycline-rifampicin (86%) compared to the other antibiotic combinations (average 69%). However, because of the retrospective study design the validity of the results is limited. A randomized clinical study is necessary to determine if doxycycline-rifampicin is superior to other conventional treatment regimens. The Dutch guideline recommends both doxycycline-rifampicin and trimethoprim-rifampicin as first choice treatments for decolonization of complicated MRSA carriage. Therefore trimethoprim-rifampicin will be the comparator of this study.

Objective: To determine the superiority of doxycycline-rifampicin compared to trimethoprim-rifampicin for the decolonization treatment of complicated MRSA carriership.

Study design: Multicenter open-label cluster randomized controlled trial.

Study population: Adult (>18 years) patients with complicated MRSA carriership, treated at one of the participating outpatient clinics. Sample size 211 patients.

Intervention: Group A: doxycycline 200 mg q.d. - rifampicin 600mg b.i.d. versus Group B: trimethoprim 200mg b.i.d. - rifampicin 600mg b.i.d. All orally, total duration 7 days.

Main study parameters/endpoints: The main study endpoint is the success rate of MRSA decolonization. Successful decolonization is defined as 3 consecutive negative cultures after treatment, with a minimum interval of 7 days.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: MRSA decolonization treatment is already standard clinical practice in the Netherlands. There is no additional burden or risk associated with participation in the study. Both antibiotic regimens (in Group A and Group B) used in the study, are recommended as first-line therapy by the Dutch guideline for the treatment of MRSA carriage. The study is open label, so there is no additional risk of blinding. The number of outpatient visits and follow-up cultures are not different from daily clinical practice in the Netherlands. No invasive procedures will be performed for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Complicated MRSA carriership. Complicated carriership is defined as having one of the following features: (i) the presence of MRSA located at another site than the nose, (ii) an active infection with MRSA, (iii) in vitro resistance for mupirocin, (iv) active skin lesions, (v) foreign material that connects an internal body site with the outside (e.g., urine catheter, external fixation material), (vi) previously failure of decolonization treatment.

In case of none of the previously mentioned features, this is considered uncomplicated carriership.

- The ability to provide informed consent for the use of their data.

Exclusion Criteria:

* - Presence of any iv-access, urinary catheters or drains (because of high risk of treatment failure)
* Failure of previous decolonization attempt of complicated MRSA carriage
* Allergy or other contra-indication to either doxycycline, rifampicin or trimethoprim (these patients will participate in the observational arm)
* Previous participation in this study (every patient can only participate once)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
success rate | 3 consecutive negative cultures after treatment, with a minimum interval of 7 days.
  success rate of MRSA decolonization

SECONDARY OUTCOMES:
long term success rate | 1 year
  success rate of decolonization treatment after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Merel Lambregts, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- LUMC, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided